CLINICAL TRIAL: NCT07169773
Title: Comparison Between Convective Radiofrequency Water Vapor Thermal Ablation (REZUM) Versus Tamsulosin in Management of Lower Urinary Tract Symptoms in Patients With Benign Prostatic Enlargement
Brief Title: Comparative Study Between Rezum and Tamsulosin
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: khaled Abdelsattar Gad Ibrahim (Other)
Responsible Party: Sponsor-Investigator, khaled Abdelsattar Gad Ibrahim, consultatnt doctor, Armed Forces College of Medicine, Cairo, Egypt
Organization: Armed Forces College of Medicine, Cairo, Egypt (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Rezum procedure for BPH
Record Dates: First submitted 2025-09-04; First posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Prostate Hyperplasia
Keywords: Rezum; tamsulosin
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Tamsulosin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rezum group (Active Comparator): 47 patient underwent Rezum therapy
  Interventions: Device: Rezum
- tamsulosin group (Active Comparator): 47 patients were given Tamsulosin medical treatment
  Interventions: Drug: Tamsulosin

INTERVENTIONS:
Device: Rezum — Rezum procedure in Rezum group
  Arms: Rezum group
Drug: Tamsulosin — Tamsulosin were given to Tamsulosin group
  Arms: tamsulosin group

SUMMARY:
the investigators aimed to compare the efficacy and safety of Rezūm therapy for the management of benign prostatic hyperplasia (BPH) with Tamsulosin.

DETAILED DESCRIPTION:
So far, data from available studies point towards good clinical outcomes with a short-term risk of self-limiting minor complications. Its application has demonstrated clinical effectiveness and possesses specific benefits that distinguish it among other treatments. It is applicable to outpatient setting, is effective in preserving sexual function and is versatile in its ability to treat a variety of prostate gland morphology.

ELIGIBILITY:
Inclusion Criteria:

1. with prostate volumes of 30- 80 mL,
2. mild to mod LUTS
3. (maximum urinary flow rate [Q max] of <15 mL/s
4. International Prostate Symptom Score [IPSS] of >13)
5. PVR urine < 250 ml

Exclusion Criteria:

1. prostate cancer,
2. neurogenic bladder
3. urethral stricture,
4. urinary bladder stone
5. previous prostatic surgery

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 94 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
The International Prostate Symptom score (IPSS) | Time Frame: for each case in both groups the investigator assess IPSS at 3, 6, 12 after procedures through study completion, an average of 1 year
  Measurement of The International Prostate Symptom score (IPSS) in both groups After 3, 6, 12 months of operation, the questioner is performed. Minimum :0 / Maximum : 35 Total score: 0-7 Mildly symptomatic; 8-19 moderately symptomatic; 20-35 severely symptomatic
The Maximum Urinary flow rate (Qmax) | Time Frame: for each case in both groups the investigator assess Qmax at 3, 6, 12 months after procedures through study completion, an average of 1year
  Measurement of The Maximum Urinary flow rate (Qmax) in both groups After 3, 6, 12 months of operation, the procedure is performed. Qmax is measured by (ml/sec) Normal values are described as a Qmax above 15 ml/sec and below 10 ml/sec is considered abnormal
The Quality of Life (QoL) | [Time Frame: for each case in both groups the investigator assess QoL at 3, 6, 12 months after procedures through study completion, an average of 1 year
  Measurement of The Quality of Life (QoL) in both groups After 3, 6, 12 months of operation, the questioner is performed. Minimum :0 means delighted / Maximum : 5 means unhappy
The Prostate size | Time Frame: for each case in both groups the investigator assess prostate size at 3, 6, 12 months after procedures through study completion, an average of 1 year.
  the prostate size was measured by grams by Trans-rectal ultra sound

SECONDARY OUTCOMES:
Incidence of complications | through 1 year
  For each case in both groups the investigator assess the safety using incidence of complications by The Clavien-Dindo system. It uses a 5-grade scale (I-V), to classify complications from minor issues not requiring intervention (Grade I) to death (Grade V).

CONTACTS AND LOCATIONS:
Locations (1):
- The Armed Forces College of Medicine (AFCM, Cairo, Nozha, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Samir M, Mahmoud MA, Abdelmonem HA, Elrefaie M, Gad KA. A comparative analysis of the outcomes of Rezum therapy based on prostate size: a four-year retrospective analysis. World J Urol. 2025 Jul 17;43(1):443. doi: 10.1007/s00345-025-05793-0. PMID 40676194
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/40676194/